CLINICAL TRIAL: NCT01670058
Title: Pattern Of Use Of Belatacept In US Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM103-074
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Kidney Transplantation: Transplantation, Kidney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Belatacept treated adult kidney-only transplant recipients: All adult kidney-only transplant recipients treated with Nulojix (Belatacept)
- CNIs at transplantation

SUMMARY:
* The prevalence of Belatacept use
* The characteristics of Belatacept users and the temporal trends in these characteristics
* Characteristics of adult kidney-only transplant recipients who are treated with Belatacept vs. who are treated with Calcineurin inhibitors (CNI)-based regimens at the time of transplantation, and the temporal trends in these characteristics during 7 years post approval of Belatacept.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* The cohort for the analyses of all transplants includes all organ transplant recipients who are reported with Belatacept at transplant

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort for the analyses of all transplants includes all organ transplant recipients who are reported with Belatacept at transplant
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of Belatacept use | Up to 72 months
  Timeframe: Every 6 months up to 72 months
Characteristics of Belatacept users, in terms of age, sex, ethnicity, transplanted organs, donor EBV infection-recipient EBV serostatus, donor CMV infection-recipient CMV serostatus, and the temporal trends in these characteristics | Up to 72 months
  EBV = Epstein-Barr virus; CMV = cytomegalovirus; Timeframe: Every 6 months up to 72 months
Characteristics of adult kidney-only transplant recipients who are treated with Belatacept vs. who are treated with CNI-based regimens at the time of transplantation and temporal trends in these characteristics during 7 years post approval of Belatacept | Up to 72 months
  Characteristics of adult kidney-only transplant recipients assessed are age, sex, ethnicity, EBV serostatus, CMV serostatus, organ characteristics, concomitant immunosuppressive medication use, and type of induction medication use.
  CNI = calcineurin inhibitors; Timeframe: Every 6 months up to 72 months

SECONDARY OUTCOMES:
Characteristics of adult EBV seropositive kidney-only transplant recipients treated with Belatacept vs who are treated with CNI-based regimens at time of transplantation & temporal trends in these characteristics during 7 yrs post approval of Belatacept | Every 6 months up to 72 months
  Characteristics of adult, EBV seropositive, kidney-only transplant recipients assessed are age, sex, ethnicity, CMV serostatus, organ characteristics, concomitant immunosuppressive medication use, and type of induction medication use
Extent of switches to or from Belatacept within one year post-transplant in adult, kidney-only transplant recipients | Every 6 months up to 72 months
Characteristics of switchers vs. non-switchers (age, sex, ethnicity, EBV serostatus, CMV serostatus, organ characteristics, concomitant immunosuppressive medication use, and type of induction medication use) | Every 6 months up to 72 months
Temporal trend in switches during 7 years post-approval | Every 6 months up to 72 months
CMV treatment/prophylaxis by CMV serostatus in adult kidney-only transplant recipients who had anti-CMV therapy data recorded in United Network for Organ Sharing (UNOS) and treated with Belatacept vs. CNIs at transplantation | Every 6 months up to 72 months
CMV treatment/prophylaxis by CMV serostatus in adult kidney-only transplant recipients who had anti-CMV therapy data recorded in UNOS and switched to Belatacept, switched from Belatacept, or did not switch | Every 6 months up to 72 months
Characteristics of Belatacept users stratified by EBV serostatus, including age, sex, ethnicity, general medical factors, transplant history (organ, date, graft failure date), and donor organ characteristics | Every 6 months up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Cherikh WS, Kou TD, Foutz J, Baker TJ, Gomez-Caminero A. Patterns of belatacept use and risk of post-transplant lymphoproliferative disorder in US kidney transplant recipients: An analysis of the Organ Procurement and Transplantation Network database. PLoS One. 2025 Jan 10;20(1):e0311935. doi: 10.1371/journal.pone.0311935. eCollection 2025. PMID 39792912
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx